CLINICAL TRIAL: NCT06202313
Title: A Multicenter, Randomized, Controlled, Open Label Clinical Study on the Treatment of Recurrent or Metastatic Triple Negative Breast Cancer With Cadonilimab Combined With Eribulin Versus Eribulin Alone
Brief Title: Study of Cadonilimab (AK104) Plus Eribulin vs. Eribulin Monotherapy for Recurrent or Metastatic Triple-negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Postdoctoral, Chief Physician, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-007
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cadonilimab + Eribulin (Experimental): Participants receive Cadonilimab 10mg/kg IV on Day 1 of each 21-day cycle PLUS Eribulin 1.4mg/m^2 IV on Days 1 and 8 of each 21-day cycle.
  Interventions: Biological: Cadonilimab; Drug: Eribulin
- Eribulin (Active Comparator): Participants receive Eribulin 1.4mg/m^2 IV on Days 1 and 8 of each 21-day cycle.
  Interventions: Drug: Eribulin

INTERVENTIONS:
Biological: Cadonilimab — Participants receive Cadonilimab 10mg/kg IV on Day 1 of each 21-day cycle PLUS Eribulin 1.4mg/m^2 IV on Days 1 and 8 of each 21-day cycle.
  Other Names: AK104
  Arms: Cadonilimab + Eribulin
Drug: Eribulin — Participants receive Eribulin 1.4mg/m^2 IV on Days 1 and 8 of each 21-day cycle.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Cadonilimab (AK104) plus Eribulin compared to the efficacy and safety of Eribulin monotherapy in the treatment of adult patients with recurrent, or metastatic triple negative breast cancer.

The primary study hypothes is that the combination of Cadonilimab (AK104) plus Eribulin is superior to Eribulin monotherapy with respect to Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as assessed by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign a written informed consent form, which must be signed before the designated research procedures required for the study are carried out.
2. Age at the time of signing the Informed Consent Form (ICF) is ≥ 18 years old and ≤ 75 years old, both male and female.
3. The Eastern Cancer Collaborative Organization (ECOG) has a physical fitness score of 0 or 1.
4. The expected survival period is ≥ 3 months.
5. Recurrent or metastatic incurable triple negative breast cancer confirmed by histology and/or cytology.
6. Having received ≤ 2-line systematic treatment for recurrent or metastatic diseases, including: ① untreated after recurrence or metastasis, but receiving paclitaxel and anthracycline drugs within 12 months before recurrence or metastasis (including neoadjuvant treatment stage and adjuvant treatment stage), Or ② After recurrence or metastasis, the subject has received 1-2 lines of treatment (including at least one anthracycline and one paclitaxel in the previous adjuvant treatment stage, neoadjuvant treatment stage, or treatment after recurrence/metastasis).
7. According to the RECIST v1.1 standard, there is at least one measurable tumor lesion. Agree to provide archived or freshly obtained tumor tissue samples (formalin fixed paraffin embedded [FFPE] tissue wax blocks or at least 5 unstained tumor tissue slice samples) to confirm PD-L1 expression.
8. The time interval between the last treatment: (a) If the last treatment is targeted therapy such as Olaparib, the interval should be ≥ 2 weeks; (b) If the last treatment is chemotherapy, an interval of ≥ 4 weeks is required.
9. Having good organ function:

   1. Blood routine examination (no blood components or cell growth factors were used to support treatment within the first 2 weeks of randomization):

      Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;

      · Platelet count ≥ 100 × 10^9/L; Hemoglobin ≥ 9.0g/dL.
   2. Kidney:

      Creatinine < 1.5 × ULN, or creatinine clearance rate * (CrCl) calculated value ≥ 50mL/min;

      *The Cockcroft Fault formula will be used to calculate CrCl: CrCL (mL/min)={(140 age) × Body weight (kg) × F} /(SCr (mg/dL) × 72) Among them: F=1 for males and F=0.85 for females; SCr=serum creatinine. Urinary protein<2+or 24-hour urine protein quantification<1.0g.
   3. Liver:

      Serum total bilirubin (TBiL) ≤ 1.5 × ULN; AST and ALT ≤ 2.5 × ULN (AST and ALT ≤ 5 for subjects with liver metastasis) × ULN, but not accompanied by elevated bilirubin); Serum albumin (ALB) ≥ 28g/L.
   4. Coagulation function:

   International standardized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN
10. Female subjects with fertility must undergo a serum pregnancy test within 72 hours before the first medication, and the result should be negative. If a female subject with fertility engages in sexual activity with an unsterilized male partner, the subject must adopt an acceptable contraceptive method starting from screening and must agree to continue using the contraceptive method for 120 days after the last dose of the study drug; Periodic abstinence and safe period contraception are unacceptable contraceptive methods. Whether to stop contraception after this time point should be discussed with researchers.

    1. Women with fertility refer to those who have not undergone surgical sterilization (i.e. bilateral fallopian tube ligation, bilateral oophorectomy, or total hysterectomy) or those who have not undergone menopause (defined as those who have ceased menstruation for at least 12 consecutive months without alternative medical reasons, and whose serum follicle stimulating hormone levels are within the laboratory reference range of postmenopausal women);
    2. An efficient contraceptive method refers to a contraceptive method with a low failure rate (such as less than 1% per year) under continuous and correct use. Not all contraceptive methods are efficient. In addition to barrier contraception, female subjects with fertility can also use hormonal contraception (such as birth control pills), intrauterine device contraception, etc. to ensure that pregnancy does not occur.

Exclusion Criteria:

1. human epidermal growth factor receptor 2 (HER2) is positive and/or hormone receptor is positive.
2. Previously received treatment with PD-1 monoclonal antibody, PD-L1 monoclonal antibody, or CTLA-4 monoclonal antibody.
3. Received systematic anti-tumor therapy within the first 4 weeks of randomization, including chemotherapy, radiation therapy, immunotherapy, targeted therapy (small molecule targeted therapy within the first 2 weeks of randomization), biological agent therapy, etc; Palliative local treatment within the first 2 weeks of randomization; Received systemic non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, etc.) within the first 2 weeks of randomization; In the first 2 weeks of randomization, they received Chinese herbal medicine or traditional Chinese patent medicines and simple preparations with anti-tumor indications.
4. Currently participating in another clinical study, unless it is an observational, non-interventional clinical study, or a follow-up period of an intervention study.
5. Have active or untreated brain metastases, meningeal metastases, spinal cord compression, or leptomeningeal diseases. However, participants who meet the following requirements and have measurable lesions outside the central nervous system are allowed to be enrolled: asymptomatic after treatment, imageologically stable for at least 4 weeks before the start of study treatment (if there are no new or expanded brain metastases), and have stopped systemic glucocorticoid and anticonvulsant drug treatment for at least 2 weeks.
6. Have clinical symptoms of pleural effusion, pericardial effusion, or pleural/ascites that require frequent drainage (≥ once per month).
7. Active autoimmune diseases that require systematic treatment within the first 2 years of randomization, or autoimmune diseases that the researcher determines may recur or plan treatment. Except for the following:

   1. Skin diseases that do not require systematic treatment (such as vitiligo, alopecia, psoriasis, or eczema);
   2. Hypothyroidism caused by autoimmune thyroiditis requires only stable doses of hormone replacement therapy;
   3. Type I diabetes requiring only a stable dose of insulin replacement therapy;
   4. Childhood asthma has completely relieved, and no intervention is required in adulthood;
   5. Researchers have determined that the disease will not recur without external triggering factors.
8. Any of the following cardiovascular or cerebrovascular diseases or risk factors:

   1. Myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, acute or persistent myocardial ischemia, symptomatic heart failure (grade 2 or above according to the New York Heart Association functional classification), symptomatic or poorly controlled arrhythmia, or any arterial thromboembolism event occurred within the first 6 months of randomization.
   2. A history of deep vein thrombosis, pulmonary embolism, or other severe thromboembolism within the first 3 months of randomization.
   3. Have major vascular diseases such as aortic aneurysm, aortic dissection aneurysm, internal carotid artery stenosis that may endanger life or require surgery within 6 months.
   4. Previous history of myocarditis and cardiomyopathy.
   5. Left ventricular ejection fraction (LVEF)<50%.
9. Toxicity that has not been alleviated by previous anti-tumor therapy is defined as failure to regress to the National Cancer Institute Adverse Event General Terminology Standard (NCICTCAE v5.0) level 0 or 1, or the level specified in the inclusion/exclusion criteria, except for hair loss/pigmentation. Subjects who have experienced ≥ 3 levels of immune related toxicity during previous treatment with immune checkpoint inhibitors are not allowed to be enrolled.

   For subjects who experience irreversible toxicity and are expected to not worsen after administration of the study drug (such as hearing loss), they may be included in the study after consultation with the medical supervisor. It is known that there are active or untreated brain metastases, meningeal metastases, spinal cord compression, or leptomeningeal diseases. However, participants who meet the following requirements and have measurable lesions outside the central nervous system are allowed to be enrolled: asymptomatic after treatment, imageologically stable for at least 4 weeks before the start of study treatment (if there are no new or expanded brain metastases), and have stopped systemic glucocorticoid and anticonvulsant drug treatment for at least 2 weeks. Subjects with long-term toxicity that cannot be restored according to the judgment of the researchers may be included in the study after consultation with medical inspectors.
10. According to the NCICTCAE v5.0 standard, it is defined as ≥ Level 2 peripheral nerve disease.
11. The presence of interstitial lung disease or non infectious pneumonia is known, and the disease is currently symptomatic or requires systemic glucocorticoid treatment in the past. Researchers have determined that it may affect the toxicity assessment or management related to the study treatment.
12. Active pulmonary tuberculosis is known to exist. Subjects suspected of active pulmonary tuberculosis need to undergo chest X-ray examination, sputum examination, and elimination through clinical symptoms and signs.
13. Received systemic anti infective therapy (excluding antiviral therapy for hepatitis B or C) within the first 2 weeks of randomization.
14. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
15. Have clinical active hemoptysis, active diverticulitis, abdominal abscess, and gastrointestinal obstruction.
16. Clinically significant bleeding symptoms or clear bleeding tendencies within the first month of randomization, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis.
17. For untreated active hepatitis B subjects (HBsAg positive and HBV-DNA more than 1000 copies/ml [200IU/ml] or higher than the lower detection limit), patients with hepatitis B are required to receive anti hepatitis B virus treatment during the study treatment period; Active hepatitis C subjects (with positive HCV antibodies and HCV-RNA levels above the detection limit).
18. Individuals with a known history of immune deficiency or HIV testing positive.
19. Known active syphilis infection.
20. Subjects who require systemic treatment with glucocorticoids (>10mg/day prednisone or equivalent dose) or other immunosuppressive drugs within the first 14 days of randomization. Except for the following:

    1. If there is no active autoimmune disease, it is allowed to use inhaled, ophthalmic, or topical corticosteroids or other corticosteroids with a dose ≤ 10mg/day of prednisone or equivalent.
    2. The dosage of systemic glucocorticoids in physiological doses is ≤ 10mg/day of prednisone or equivalent doses of other glucocorticoids.
    3. Glucocorticoids are used as pretreatment for infusion related reactions or allergic reactions (such as medication before CT examination).
21. Received live vaccine within 30 days prior to randomization, or planned to receive live vaccine during the study period.
22. A history of severe hypersensitivity to other monoclonal antibodies is known.
23. Subjects who have a known history of allergic or hypersensitive reactions to cardunizumab, iribrin, or any of their components.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator | Up to approximately 1 year
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 as assessed by Investigator will be presented.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 2 years
  OS is defined as the time from randomization to death due to any cause.
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by Investigator | Up to approximately 1 year
  ORR is defined as the percentage of the participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters).
Duration of Response (DOR) Per RECIST 1.1 as Assessed by Investigator | Up to approximately 1 year
  For participants who demonstrate CR or PR, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death. The DOR per RECIST 1.1 as assessed by Investigator will be presented.
Number of Participants Who Experience an Adverse Event (AE) | From randomization through 30 days after last dose of study treatment
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be presented.
Number of Participants Who Experience a Serious AE (SAE) | From randomization through 90 days after last dose of study treatment
  An SAE is defined as any untoward medical occurrence that, at any dose: a.) Results in death; b.) Is life-threatening; c.) Requires inpatient hospitalization or prolongation of existing hospitalization; d.) Results in persistent or significant disability/incapacity; e.) Is a congenital anomaly/birth defect; f.) Other important medical events; h.) Is a new cancer (that is not a condition of the study) or i.) Is associated with an overdose. The number of participants who experience an SAE will be presented.
Number of Participants Who Experience an Immune-related AE (irAE) | From randomization through 90 days after last dose of study treatment for serious irAEs
  AEs associated with Cadonilimab exposure may be a result of an immune response. These irAEs may occur shortly after the first dose or several months after the last dose of Cadonilimab treatment and may affect more than one body system simultaneously. For this study irAEs include, but are not limited to:
  Pneumonitis; Diarrhea/Colitis; Aspartate transaminase (AST)/Alanine transaminase (ALT) elevation or Increased bilirubin; Type 1 diabetes mellitus or Hyperglycemia; Hypophysitis; Hyperthyroidism; Hypothyroidism; Nephritis and Renal dysfunction; and Myocarditis. The number of participants who experience an irAE will be presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No